CLINICAL TRIAL: NCT07029685
Title: Effect of an Ecological Model-Based Physical Activity Intervention on Improving Obesity Parameters and Quality of Life in Preschoolers 4 to 6 Years of Age
Brief Title: Physical Activity Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrés Godoy Cumillaf (Other)
Responsible Party: Sponsor-Investigator, Andrés Godoy Cumillaf, PhD scientist, Universidad Autónoma de Chile
Organization: Universidad Autónoma de Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UAutonomaEFI; 22-25 (Other: UAUTONOMA)
Record Dates: First submitted 2025-06-04; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Healthy Children
Keywords: Physical activity; Body composition; preschool; physical fitness
MeSH Terms: conditions — Motor Activity | interventions — Restraint, Physical; Exercise

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Investigator
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one (Experimental)
  Interventions: Other: Physical
- two (No Intervention)

INTERVENTIONS:
Other: Physical — They will carry out a physical activity intervention based on the ecological model
  Other Names: Exercise
  Arms: one

SUMMARY:
Obesity is a problem that affects almost every region of the world. In Chile, data indicate that the prevalence of obesity in preschool children aged 4 to 6 years is 58%, which increases as they reach adolescence and adulthood. The role played by physical inactivity in the development of obesity is so relevant that it has been established that in children it is one of the factors that most contributes to the development of obesity. Among factors that influence adherence to healthy lifestyles are motor competence (CM) and physical condition (CF); Both CM and CF are factors that generate an underlying mechanism that decreases the risk of obesity and promotes health. Health-related quality of life [HRQoL] refers to an individual's subjective perception of the impact of health status on their physical, psychological, and social functioning. Overweight and obesity influence HRQoL. Physical activity interventions applied from an early age have proven to be a useful means of preventing childhood obesity, being more effective when implemented in the school environment and is key to achieving long-term results. The ecological model of physical activity favors modifying active lifestyle behaviors including intrapersonal, interpersonal, organizational, community, physical-environmental and political factors. Using the ecological model, physical activity interventions have managed to increase the levels of physical activity since the child and the entire environment that surrounds him or her are involved, that is, they have included the biological and behavioral, along with the motivational, school, in addition to taking into account environmental, cultural and socioeconomic aspects. The general objective of the project is to determine the effect of a physical activity intervention based on the ecological model, in the improvement of obesity parameters and quality of life in preschoolers from 4 to 6 years old. The study is experimental through a cluster-randomized clinical trial; of pre and postest.

The methodological approach is mixed. Physical Condition will be measured through the PREFIT battery with the following components:

body composition (weight, waist circumference; hip circumference, BMI); Musculoskeletal capacity (upper body strength, lower body strength; speed/agility); Cardiorespiratory capacity. Motor competence will be measured through the Children's Movement Assessment Battery (MABC-2) with the following components: Manual dexterity; Marksmanship and catch; Balance. Health-related quality of life will be assessed through the KINDL-R questionnaire for parents, in the validated version in Spanish; Sedentary behaviour and physical activity ActiGraph wGT3X-BT accelerometers will be used. To determine the effect, statistical tests will be applied for intragroup analysis and intrasubject repeated measures, considering p <.05 as significance. When statistically significant differences are found, the effect size will be calculated. In addition, the use of mixed regression models is contemplated where the models will be adjusted for baseline values and age. It is hypothesized that the physical activity intervention based on the ecological model will lead to a 3% decrease in body fat, improves anthropometric measurements, physical condition, improved competence and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

Be enrolled in the selected establishment Have the consent of the parents or legal guardian to participate in the activity Have the consent of the child when asked to participate

Exclusion Criteria:

Health impairments that limit participation in the physical activity intervention Have completed less than 80% of the intervention program

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Fat Mass | From enrollment to the end of treatment at 16 weeks
  body fat measurement
Fat Mass | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Educacion, Temuco, Chile

IPD SHARING:
Plan to Share IPD: No